CLINICAL TRIAL: NCT02372487
Title: Sildenafil Citrate Therapy for Oligohydramnios
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Hayat National Hospital (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ob/gyn 3
Record Dates: First submitted 2015-02-10; First posted 2015-02-26 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Pregnancy Complication
MeSH Terms: conditions — Pregnancy Complications | interventions — Sildenafil Citrate; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fluid therapy and sildenafil citrate (Active Comparator): Patients in first group will receive 2 liters of isotonic saline through intravenous infusion over a period of 4 hours using a rate of 250 ml per hour in addition to sildenafil citrate therapy (Viagra®) as 25 mg 3 times daily during hospitalization. After discharge patients in first group will be asked to continue sildenafil citrate therapy (Viagra®) as 25 mg 3 times daily plus a daily oral fluid intake of 2 liters
  Interventions: Drug: sildenafil citrate; Dietary Supplement: fluid therapy
- fluid therapy (Active Comparator): Patients in second group will receive 2 liters of isotonic saline through intravenous infusion over a period of 4 hours using a rate of 250 ml per hour. After discharge patients wil be asked to have 2 liters daily oral fluid
  Interventions: Dietary Supplement: fluid therapy

INTERVENTIONS:
Drug: sildenafil citrate — sildenafil citrate 25 mg every 8 hours
  Arms: fluid therapy and sildenafil citrate
Dietary Supplement: fluid therapy — 2 liters of fluid per day

SUMMARY:
The aim of this randomized trial is to detect whether or not the use of Sildenafil citrate therapy will increase the amniotic fluid volume expressed in term of amniotic fluid index measured via ultrasound for fetuses of pregnancies complicated by oligohydramnios, and to compare the outcomes of Sildenafil-treated pregnancies with similar pregnancies that will remain Sildenafil-naïve.

DETAILED DESCRIPTION:
Women who will be referred to the maternity ward of both hospitals for a checkup and have the inclusion criteria will be offered admission for at least 24 hours to have complete rest aiming to increase the placental blood circulation of the uterus, which by itself can improve the amniotic fluid level. Patients will be randomly allocated into two groups according to a trial sequence determined via a computer generated random table. The trial sequence is hidden into opaque sequenced envelopes as each envelope contains an assignment for a single patient. Patients in first group will receive 2 liters of isotonic saline through intravenous infusion over a period of 4 hours using a rate of 250 ml per hour in addition to sildenafil citrate therapy (Viagra®) as 25 mg 3 times daily and the same fluid regimen will be used in control group but without sildenafil citrate treatment. During hospital course maternal monitoring will be done using maternal vital signs for early detection of any manifestations of fluid overload while fetal monitoring will be done using non-stress test and all patients less than 34 completed weeks will receive dexamethasone in a total dose of 24mg to enhance fetal lung maturity in case expedited delivery is needed. Fasting will also be recommended during fluid therapy in case any emergency interference is required then all patients will resume their usual daily diet and fluid intake. All patients will then undergo sonography after 24 hours for reassessment of amniotic fluid index and those who will show an improvement of at least 20% will be discharged home and for those who still show no results the same regimen will be repeated. Discharged patients in first group will be asked to continue sildenafil citrate therapy (Viagra®) as 25 mg 3 times daily plus a daily oral fluid intake of 2 liters while those in the control group will be asked only to have 2 liters daily oral fluid. Outpatient monitoring in both groups will depend on twice weekly non-stress test and once weekly amniotic fluid index and biophysical profile. Readmission and inpatient therapy using same protocol in each group will be indicated at any time if amniotic fluid index reduced to ≤ 5 cm. All patients also will be instructed to undergo periods of bed rest and, also they will be educated to count fetal kicks and to report immediately to the hospital if being unsatisfactory.

Patients in both groups will be monitored till they will go into spontaneous labor or till delivery will be indicated. The primary outcome measure will be the values of amniotic fluid index before and after therapy in each group and between both groups. The secondary outcome measures will be mode of delivery, gestational age at birth, fetal birth weight, and fetal and neonatal outcomes (Apgar scores, umbilical artery acid-base analysis at birth, and the need for transfer to the neonatal intensive care unit) which will be analyzed for the study and control groups.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women will be included if they are of:

1. any age, any parity
2. carrying a singleton pregnancy
3. gestational age (GA) 30 weeks or more (based on the last menstrual period and confirmed by the results of ultrasound or determined through early pregnancy sonography)
4. Amniotic fluid index ≤ 5
5. no pregnancy complications such as preeclampsia, gestational hypertension, or diabetes
6. no prior history of kidney, lung, and heart disease (the use of bolus-fluid therapy is contraindicated in these patients)
7. intact fetal membranes.

Exclusion Criteria:

1. Mothers treated with prostaglandin synthetase inhibitors
2. well established labor
3. evidence of fetal distress (non-reactive non stress test)
4. fetal complications (intrauterine growth retardation or obvious fetal anomalies)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
the values of amniotic fluid index before and after therapy in each group and between both groups | 9 months

SECONDARY OUTCOMES:
mode of delivery | 9 months
gestational age at birth | 9 months
fetal birth weight | 9 months
Apgar scores | 9 months
the need for transfer to the neonatal intensive care unit | 9 months

CONTACTS AND LOCATIONS:
Locations (2):
- Menoufia University, Shebin Elkom, Egypt
- Alhayah national hospital, Abhā, Saudi Arabia

REFERENCES:
- [Derived] Maher MA, Sayyed TM, Elkhouly N. Sildenafil Citrate Therapy for Oligohydramnios: A Randomized Controlled Trial. Obstet Gynecol. 2017 Apr;129(4):615-620. doi: 10.1097/AOG.0000000000001928. PMID 28277352 (Retraction: PMID 32150003 Obstet Gynecol. 2020 Apr;135(4):980)